CLINICAL TRIAL: NCT06585722
Title: The Association Between Venous Excess Ultrasound, the Lung Ultrasound Score and Acute Kidney Injury and Death in the Intensive Care Unit Population
Brief Title: Association Between Venous Excess Ultrasound Grading System and Acute Kidney Injury in the ICU Population
Acronym: VExUS ICU
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, P.R. Tuinman, Dr. P.R. Tuinman, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2020.01111
Record Dates: First submitted 2024-03-13; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Fluid Overload; Kidney Injury; Make-30
MeSH Terms: conditions — Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Fluid resuscitation is one of the cornerstones of treatment in ICU patients. Nonetheless, excessive fluid administration can lead to fluid overload which has been associated with worse outcomes in the ICU. To prevent this, assessments of fluid responsiveness are commonly employed. However, fluid responsiveness does not take fluid tolerance into account. Fluid tolerance is the idea that a patient might still be fluid responsive but might already be at risk of the detrimental effects of fluid therapy. Recent developments in point of care ultrasound e.g. the Venous excess ultrasound might help identify patients at risk of fluid overload. However its association with patient relevant outcomes in the ICU remains unclear.

DETAILED DESCRIPTION:
This study will investigate the association between the venous excess ultrasound grading system (VExUS) and patient relevant outcomes such as acute kidney injury, mortality and length of stay.

A secondary analysis is planned where the association between VExUS and the lung ultrasound score will be investigated

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU 18 years or older expected to stay in the ICU for more than 24 hours

Exclusion Criteria:

* any obstruction between the righ atrium and structures assessed by VExUS
* a medical history of: Major cardiac shunts (e.g. atrial septum defect), Tricuspid regurgitation, dialysis, portal hypertension, pulmonary hypertension, interstitial lung disease, recipients of a kidney of liver transplant.
* patients in whom an ultrasound assesment is unfeasible e.g. a BMI over 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cricitally ill patients who are expected to be admitted to the ICU for more than 24 hours and who do not meet the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09-05 (Estimated); Study Completion 2024-09-05 (Estimated)

PRIMARY OUTCOMES:
Rate of acute kidney injury | within 30 days of admission to the ICU
  Clinically relevant acute kidney injury in the ICU: a 200% rise in creatinine or the use of renal replacement therapy
Mortality | within 30 days of admission to the ICU
  death of all causes
Rate of MAKE-30 | within 30 days of admission to the ICU
  a composite endpoint of mortality and acute kidney injury ( including renal replacement therapy)

OTHER OUTCOMES:
Lung ultrasound score | maximum of 3 times during the first 7 days of admission
  a score for lung aeration as assessed by ultrasound ranging from 0 to 36 where 0 is the normal physiological state
Cardiac function as assed by ultrasound | maximum of 3 times during the first 7 days of admission
  determined by eyeballing and measurement of the tricuspid annular plane systolic excursion (>16 is normal)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided